# **Cover Page to Accompany ClinicalTrials.gov Document**

#### **Informed Consent**

for

Pilot Study of the Physiological Effects of an Integrative Medicine Approach in Irritable Bowel Syndrome

June 6, 2019

Thomas Jefferson University IRB ID: 17D.184

**Clinical Trial Number: NCT03370614** 

Thomas Jefferson University **Informed Consent Document for Human Subjects Research** 

Department: Emergency Medicine and Radiology Principal Investigator: Andrew B. Newberg, MD Telephone: 215-503-3422 Co -Investigator: Daniel A. Monti, MD **Telephone**: 215-955-4410 Medical Study Title: Pilot Study of the Physiological Effects of an Integrative Medicine Approach in Irritable Bowel Syndrome Lay Study Title: PET-MRI in IBS

#### What Is Informed Consent?

1

2

3 4

5 6

7 8

9

10 11

12 13

14 15

16

17

18

19 20

21 22

23 24

25

26

27 28

29 30

31

32

33

34

35 36 37

38

39

40

41

42

43

You are being asked to take part in a medical research study. As required by federal regulations, this research study has been reviewed and approved by an Institutional Review Board (IRB), a University committee that reviews, approves and monitors research involving humans. Before you can make a knowledgeable decision about whether to participate, you should understand the possible risks and benefits related to this study. This process of learning and thinking about a study before you make a decision is known as informed consent and includes:

• Receiving detailed information about this research study:

- Being asked to read, sign and date this consent form, once you understand the study and have decided to participate. If you don't understand something about the study or if you have questions, you should ask for an explanation before signing this form;
- Being given a copy of the signed and dated consent form to keep for your own records.

You should understand that your relationship with the study doctor is different than your relationship with your treating or personal doctor. The treating doctor treats a specific health problem with the goal of improving a medical condition. A study doctor treats all subjects according to a research plan to obtain information about the experimental drug, device or procedure being studied and with the understanding that you may or may not benefit from being in the study. You should ask questions of the study doctor if you want to know more about this.

#### What is the purpose of this study?

You have symptoms of Irritable Bowel Syndrome which means that you have experienced significant gastrointestinal (GI) symptoms. It is important to understand the brain and GI mechanisms of IBS in order to better determine therapeutic interventions to reduce pain. Part of the difficulty in treating IBS is to determine how better to diagnose what specific issues are affecting the brain and GI tract that result in symptoms. In order to assess the brain and GI tract

Approval Date 3/11/2/ Expiration Date 3/11/22

PET-MRI IBS OHR-8 2017 08 17REV 2019 05 14 rev 2019 06 6b

Annual review due 6 weeks before expiration.

function more effectively, we would like to have you undergo a small battery of diagnostic tests that include magnetic resonance imaging (MRI), positron emission tomography (PET). In addition, you will receive several questionnaires and a clinical evaluation to determine the nature and level of your IBS symptoms. A secondary goal of this study is to determine if integrative therapy based on diet and nutritional counseling will improve your IBS symptoms and alters GI or brain physiology. All subjects will receive the dietary and nutritional counseling program. The dietary and nutritional counseling will begin with a one hour session to review the diet and nutrition program in detail. We will contact you a minimum of once a month to review the recommendations, answer any questions you have, and help ensure that you are following the dietary recommendations. Prior to starting this intervention and at the end of approximately 2 months of receiving it, you will undergo the brain and body scan evaluation and receive clinical and pain testing. 

# How many individuals will participate in the study and how long will the study last?

We hope to enroll up to 60 patients at Jefferson. The entire study will take about 2 years to complete. Your involvement in the study will last about 3 months.

#### What will I have to do during the study?

The informed consent process will be completed with you. You will be asked questions about your medical history and about the medications you are taking. You will also be asked to complete several questionnaires about your mood, quality of life, and your GI symptoms which will take no longer than one hour to complete. You will also undergo a clinical examination evaluating your GI symptoms in order to determine how much they affect you. A full set of laboratory values will be obtained including measures of inflammation. You will repeat this process including the questionnaires and examination again in 2 months. You may also undergo an initial stool analysis. Throughout the study, you will continue to take whatever medications your doctor has prescribed for you. However, we will ask you to try to remain at the same dosage of any medication throughout the study unless your doctor changes the dose because of worsening symptoms or because of side effects.

You will initially receive two different scans that will be performed simultaneously in a special combined scanner. One scan, called positron emission tomography (PET), will evaluate your brain and body metabolism to determine which areas of your brain and which parts of your body are functioning differently. The other scan, called magnetic resonance imaging (MRI) will evaluate the structure and function of the brain, along with the connecting fibers affected by pain. On the day of both scans, you will report to the Marcus Institute of Integrative Health at 789 E. Lancaster Avenue in Villanova, PA 19085.

Thomas Jefferson University
Andrew Newberg, MD
PET-MRI in IBS
215-503-3422
IRB Control 17D.184
Page 3 of 9

Female subjects of child bearing potential will first have a pregnancy test and if negative will proceed with the remainder of the study. The PET scan measures the energy metabolism in the brain and body which is particularly affected by pain symptoms. The PET scan works by injecting into your vein a radioactive medicine called FDG. FDG is a form of the sugar, glucose that is used by your brain for energy. By injecting the FDG, we can see where in the brain and body it goes so that we can take a picture of the activity in these areas. After injection of the tracer, you will be asked to rest quietly in a dimly lit room for approximately 30 minutes. At that point, you will be brought into the scanner room and will lie down on the PET imaging table. The remainder of the procedure involves having your head held comfortably in a special head holder as a reminder not to move your head and remain still while the scanner takes pictures of your brain. Immediately after the brain scan, you will be allowed to have a brief break (no more than 5 minutes) and then we will scan your abdomen and pelvis (to see your GI tract).

The MRI scan is performed simultaneously with the PET scan using a special PET-MRI scanner that can do both at the same time. Before the MRI scan, we will ask you a number of questions to make sure you do not have any metal in your body that might affect the scanner. The MRI scans add no radiation, but do make loud banging noises for which you will be given ear plugs to block the sound. The MRI, along with the PET scan, is done over a total period of time of about 60 minutes.

After you receive the initial diagnostic testing above, you will receive the dietary and nutritional counseling which will last approximately one hour. This program will be individualized to your specific dietary/nutrition problems as they are related to your IBS. In addition, we will contact you in one month by phone (or in person if you desire) to answer questions and help ensure that you are following the diet and nutrition recommendations. After following the dietary/nutrition program for two months, you will return for your follow up visit in which you will undergo the same imaging and diagnostic testing as you did initially. That will conclude your participation in the study.

#### What are the risks or discomforts involved?

## Integrative Dietary and Nutritional Counseling Program

The diet is a healthful diet that provides all the essential dietary requirements. Anytime a diet is changed, gastrointestinal discomfort or symptoms may occur.

#### PET Risks

Use of FDG PET imaging is commercially approved, and has resulted in very rare adverse effects of skin redness, facial swelling, fever, and short lasting rise in blood pressure. This research study involves exposure to radiation from the FDG PET scan and therefore you will receive a radiation dose that you would not receive if you did not have the scans. The radiation dose obtained as the result of participating in this study is the same as standard clinical brain scans using the same tracers. Therefore, at the doses you will receive, it is very likely that you will see no effects at all. Please inform the investigator of any participation in previous studies involving radiation exposure. Cumulative radiation doses have been associated with some forms *PET-MRI in IBS 2017 08 17 REV 2019 05 14 rev 2019 06 06b* 

- of cancer, and thus, repeated exposure to radiation should be minimized. The radiation exposure
- from the FDG PET scan is equivalent to flying in an airplane across the country. Some persons
- may experience some discomfort while lying flat on the table for the PET-MRI scan or may feel
- uncomfortable or anxious in the scanner. Subjects may feel hungry, dizzy or light-headed from
- fasting prior to the FDG scan. Since the injection of the FDG requires inserting a needle into
- your arm vein, there can be pain and discomfort at the injection site. Bleeding and infection may
- also occur.

136

- 137 MRI Risks
- 138 You will be asked to complete a MRI Patient Information History form. The MRI scan does not
- involve any radiation exposure. Due to the strength of the magnetic field of the MRI, there is a
- risk of being injured if an unsecured metal object flies into the MRI scanner. In order to
- minimize this risk, you will be asked to remove all metal objects from your person. Also, all
- metal objects will be cleared from the area prior to the scan. This is the standard practice when
- patients undergo MRI exams. It is important when discussing the study that you inform the staff
- if you have any of the following:
- 145 Surgically implanted electrical devices
- 146 Pacemaker
- 147 Surgically placed metallic clips (aneurysm clips)
- 148 Ear implants
- 149 Any history of metal fragments in the eye

150151

Some persons may experience some discomfort while lying flat on the table for MRS scans or may feel uncomfortable or anxious in the scanner.

152153154

- Survey Question and Clinical Examination Risks
- Some of the questions we will ask you as part of this study, as well as the neurological
- examination, might make you feel uncomfortable. You can refuse to answer any of the questions
- and you are free to take a brief break at any time when answering these questions or while
- undergoing the clinical exam. However, you must complete the questionnaire or clinical exam
- during the study period.

160 161

- Risks of Discovering an Incidental Finding
- The result of the scans will be reported in a clinical report by a trained specialist. If an unknown
- abnormality (also called an incidental finding) is discovered on the PET or MRI scan, you will be
- thoroughly counseled by the study doctor and will have an opportunity to ask any questions.
- Such a finding may make you feel anxious or depressed. However, the information and scans
- will be made available to your primary care doctor or referring physician in order to manage the
- finding as quickly and effectively as possible.

168

- 169 What To Do If You Experience Any Adverse Effects
- You should call the study doctor as soon as possible at 215-503-3422 if, during the course of this
- study, you develop any side effects or symptoms. The study doctor has told you that if your
- 172 condition worsens, if side effects become very severe, or if it turns out that being in this study is
- not in your best interest, you will be taken out of the study.

PET-MRI in IBS 2017 08 17 REV 2019 05 14 rev 2019 06 06b

## What are the risks to fetuses, infants and pregnant women?

Pregnant women or women who are breast feeding should not be in this study because exposure to the radioactive materials may be hazardous to an embryo, fetus or nursing infant. Even medications that are well known and prescribed may have adverse effects on an embryo or fetus. Since this study also includes radiation related to the FDG PET scans, pregnant women or women who are breast feeding should not be in this study. As with any medication, there are unknown risks. To be in this study you and your partner must practice adequate birth control measures. The study doctor will discuss acceptable methods of birth control with you. If you are a woman of childbearing potential, you will have a pregnancy test before making a decision about being in this study. This requires either a urine test or that blood be drawn from a vein in your arm (1-2 tsp.) one or two days prior to the start of the study. The results of this pregnancy test will be made available to you prior to the start of the study.

If you become pregnant during the course of this study, you should notify the study doctor as soon as possible.

If you are a person in a same sex relationship, it is not necessary for you to practice birth control. However, if you are female, you will still have to have pregnancy tests according to the study protocol.

#### Are there alternatives to being in the study?

You do not have to participate in this study.

# How will privacy and confidentiality (identity) be protected? Federal regulations require that certain information about individuals be kept confidential. This

information is called "protected health information" (PHI). PHI includes information that identifies you personally such as name, address and social security number, or any medical or mental health record, or test result, that may have this sort of information on it. The laws state that you may see and review your TJU or Thomas Jefferson University Hospital medical records at any time. However, in a research study, you may not see the study results or other data about the study until after the research is completed unless the study doctor decides otherwise.

If you join this study, the following individuals or entities may have access to your PHI and by law must protect it. These include investigators listed on this consent form and other personnel of Thomas Jefferson University and Thomas Jefferson University Hospitals, Inc. involved in this specific study, the University's Division of Human Subjects Protection and the Institutional Review Board (IRB), and your health insurance company (if necessary for billing for standard medical care).

Your PHI may also be shared with the following entities that, while not obligated by law to protect PHI, will protect it to the best of their ability:

- The Principal Investigator or designate, who will oversee the study and review medical records to ensure study-related information is correct,
- With any person or agency required by law.

If you develop an illness or injury during the course of your participation in this study, other PHI about treating and following the condition may be generated and disclosed as it relates to this study. Your PHI may be used/disclosed until the end of the research study.

You may quit the study and revoke permission to use and share your PHI at any time by contacting the principal investigator, in writing, at: Andrew Newberg, 925 Chestnut Street, Suite 120, Philadelphia, PA 19107. If you quit the study, further collection of PHI will be stopped, but PHI that has already been collected may still be used.

After the completion of the study or at the participant's request, the results of these scan will be made available to your primary care and referring physician for their clinical decision making. The results of clinical tests and procedures performed as part of this research may be included in your medical records. The information from this study may be published in scientific journals or presented at scientific meetings but you will not be personally identified in these publications and presentations.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, this Web site will include a summary of the results. You can search this Web site at any time.

## What if I am injured as a result of being in this study?

In the event that you experience a research-related injury, necessary and available medical care (including hospitalization) will be provided. A research-related injury is a physical injury or illness resulting to you that is directly caused by any procedure or treatment used in this study that is different from the treatment you would receive if you were not participating in a research study. If you are physically injured due to any drug/substance or procedure properly given under the plan for this study, the medical expenses for treating the injury will be billed to your insurance carrier. You should be aware that some costs may not be covered by insurance. There is no plan to provide compensation for loss of wages, lost time from work, personal discomfort, or for injuries or problems related to your underlying medical condition(s).

If you receive a bill related to a research-related injury that seems wrong, please discuss it with the study doctor or research coordinator.

## Will I benefit from being in this study?

You may not benefit from being in this research, but we hope that what we learn may be helpful to future patients or society in general.

Will I be paid for being in this study?

You will not receive any payment for participating in the study, but you will have access to your scans and other clinical data as well as have the opportunity to receive dietary and nutritional counseling.

#### Will I be told about any new findings?

You will be told about any new findings obtained from your diagnostic scans.

#### **Disclosure of Financial Interest**

None of the investigators has any financial interest in the companies that provide products for this study.

#### Are there costs related to being in this study?

There will be no charge to you or your health insurance for any of the PET or MRI scans, or for the dietary and nutritional counseling program as a part of this study.

If you receive a bill that you think is wrong, please discuss it with the study doctor or research coordinator.

#### **Standard Testing Procedures**

All testing procedures that are part of this research study are for research purposes only. You will not be billed for any of these procedures.

If you receive a bill that you think is wrong, please discuss it with the study doctor or research coordinator.

## Can I be removed from the study or quit the study?

Your decision to participate in this research study is entirely voluntary. You have been told what being in this study will involve, including the possible risks and benefits.

Your participation in this research project may be terminated by the study doctor without your consent/assent for any reason that he/she feels is appropriate, particularly if it pertains to your health or if you are not following the dietary/nutritional program.

You may refuse to participate in this investigation or withdraw consent and quit this study without penalty and without affecting your ability to receive medical care at Thomas Jefferson University.

If you withdraw from this study, you may continue treatment with your Jefferson doctor, or you may seek treatment from another doctor of your choice. 

Should you decide to withdraw from the study, please be sure to inform the study doctor.

Additional tests or procedures may be needed to ensure your safety. The study doctor will explain why these tests or procedures are necessary.

#### **CONTACT INFORMATION**

| Telephone number for questions | The Jefferson Institutional | 215-503-8966 |
|---|---|---|
| about your rights as a research | Review Board | |
| participant | | |
| For questions, concerns or complaints | Principal Investigator | 215-503-3422 |
| about the research, or if you suspect a | Andrew B. Newberg, MD | |
| research-related injury | | |
| | Co-Investigator, | 215-955-4410 |
| | Daniel A. Monti, MD | |
| • | Program Manager, | 215-503-3423 |
| | Nancy Wintering, LCSW | |
| If you have difficulty contacting the | Call the Jefferson Office of | 215-503-0203 |
| study staff | Human Research | |

If you want more information about the Jefferson Institutional Review Board or Jefferson's Human Research Protection Program, please visit our website at http://www.jefferson.edu/human research/irb/index.cfm

Thomas Jefferson University
Andrew Newberg, MD
PET-MRI in IBS
215-503-3422
IRB Control 17D.184
Page 9 of 9

| Non-Waiver of Legal Righ | ts Statement | |
|---|---|---|
| By your agreement to part<br>waiving any of your legal r | icipate in this study, ights. | and by signing this consent form, you are no |
| In order to be in this resear | rch study, you must | sign this consent form. |
| You affirm that you have read this consent form. You have been told that you will received | | |
| | Signatures: | |
| Your Name (please print or | type) | |
| | (Date) | (Date) |
| Your Signature | | Witness Signature |
| | | (Only required if subject understands and speak<br>English, but cannot read English, or if subject is blin<br>or cannot physically sign the consent form—delete<br>inapplicable) |
| with a description o | | s/he <b>personally</b> provided the study participan<br>rocedures, risks, benefits and alternatives to |
| participation. | | |
| Name of Person Conducting | Consent Interview | |
| | (Data) | |
| Signature of Person Conduct | (Date) ing Consent Interview | |
| | (Date) | |
| Signature of Principal Investi | igator or | |
| Co-Investigator | | |